CLINICAL TRIAL: NCT04269785
Title: Post-ablation Inflammatory Response and Endothelial Function in the Development of Early Recurrence of Atrial Tachyarrhythmia After Pulmonary Vein Isolation; Implications for Pulmonary Vein Reconnection and Freedom From Atrial Fibrillation
Brief Title: Inflammatory and Endothelial Function Response, and Arrhythmia Recurrence Following Catheter Ablation for Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Karan Saraf (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor-Investigator, Karan Saraf, Investigator, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262517
Record Dates: First submitted 2020-01-23; First posted 2020-02-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
Keywords: atrial fibrillation; ablation; radiofrequency; cryoballoon; inflammation; endothelial function; recurrence
MeSH Terms: conditions — Atrial Fibrillation; Inflammation; Recurrence | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: 20 patients with paroxysmal AF or short-lived persistent AF (less than 6 months' duration), randomised to receive ablation by radiofrequency (RF) or cryoballoon (CB) in a 1:1 allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation (Active Comparator): These patients will receive ablation by radiofrequency catheter, guided by of 3-dimensional electro-anatomic mapping technology
  Interventions: Device: Radiofrequency ablation
- Cryoballoon ablation (Active Comparator): These patients will receive ablation by cryoballoon catheter, guided by X-ray fluoroscopy
  Interventions: Device: Cryoballoon ablation

INTERVENTIONS:
Device: Cryoballoon ablation — Ablation aimed at performing pulmonary vein isolation for atrial fibrillation using cryoballoon catheter (cold therapy)
  Arms: Cryoballoon ablation
Device: Radiofrequency ablation — Ablation aimed at performing pulmonary vein isolation for atrial fibrillation using radiofrequency catheter (heat therapy)
  Arms: Radiofrequency ablation

SUMMARY:
Current international guidelines recommend a three-month blanking period after pulmonary vein isolation (PVI) for atrial fibrillation (AF). Early recurrence of atrial tachyarrhythmia (ERAT; comprising of AF, left atrial tachycardia and atrial flutter) is common, occurring in up to 65% of patients, but in the first month is generally thought not to predict long-term AF recurrence, and re-intervention is not recommended. Suggested causes for ERAT include inflammation and arrhythmogenic structural changes caused by ablation lesions. Early, purely inflammatory ERAT would not lead to late AF recurrence as pulmonary vein reconnection is established as the main factor associated with long-term recurrence in paroxysmal AF. Previous studies have shown ERAT in the second to third month (rather than first month) to be a stronger predictor of late AF recurrence, due to presumed reduction in the contribution of the acute inflammatory response after this. Biochemical data have shown that the post-ablation inflammatory phase is usually limited to the first month after both radiofrequency (RF) and cryoballoon (CB) ablation, though inflammatory markers have been shown to be less elevated following CB PVI. Histologically, lesions formed by the two modalities differ significantly. RF lesions are characterised by irregular boundaries and significant disruption to the endothelium, exposing the sub-endothelial layer and resulting in significant and sustained platelet activation, changes which can last for many months. CB lesions on the other hand, are observed as well demarcated and homogenous within one week, with reduced thrombogenicity, which may lead to reduced inflammation. ERAT following CB ablation cannot be accurately predicted by inflammatory response and it is postulated that endothelial function may play a role in the development of ERAT in such patients. Some studies have shown reduced recurrence rate and re-hospitalisation amongst the CB population, including the FIRE and ICE trial, potentially resulting in a better patient experience with CB and the possibility of a shorter blanking period. Post-ablation inflammatory response is more predictive of ERAT following RF than CB PVI, and the latter is considered to be associated with less inflammation. There is however, a paucity of data evaluating endothelial function post-AF ablation and its correlation with ERAT or late recurrences of arrhythmia. Given that earlier re-intervention in patients with ERAT in the third month of the blanking period can result in greater outcomes with respect to late recurrence of AF, if it can be demonstrated that endothelial function testing in the first few months post-CB PVI can be predictive of later ERAT, then shortening the blanking period following CB PVI and performing repeat ablation to control troublesome later ERAT may reduce overall patient morbidity and re-hospitalisation.

The purpose of this novel pilot study is to examine the relationship between the post-ablation inflammatory response, endothelial function and timing and frequency of ERAT for patients undergoing RF and CB PVI for paroxysmal or short-lived persistent (less than 6 months' duration) AF. If the initial data provides hypothesis generating information, the aim would be to perform the study on a larger basis with higher statistical power to determine whether early post-ablation endothelial function testing can predict recurrences and identify those suitable for earlier re-intervention.

ELIGIBILITY:
Inclusion criteria

* Age 18-75 years
* Paroxysmal AF or persistent AF of less than 6 months' duration
* Structurally normal heart on transthoracic echocardiogram other than mild left atrial dilatation (<34ml/m2, indexed to body surface area)
* Due to undergo pulmonary vein isolation on clinical grounds

Exclusion criteria

* Known genetic/inherited disorder that predisposes to atrial fibrillation, or Brugada syndrome
* Metabolic syndrome as defined by National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP III) criteria
* Obesity (BMI>40)
* Inability or unwillingness to receive oral anticoagulation with a vitamin K antagonist (VKA) or non-VKA oral anticoagulant (NOAC)
* Known atrial flutter
* Ischaemic heart disease documented by coronary or CT angiography, or confirmed history of myocardial infarction
* Current stage II or III hypertension (diastolic BP >100mmHg, systolic BP>160mmHg) confirmed on serial readings or ambulatory monitoring
* Diabetes mellitus other than diet controlled
* Previous catheter or surgical ablation procedure for AF
* Unwillingness or inability to complete the required follow-up arrangements
* Persistent AF > 6 months' duration or permanent AF
* Prior prosthetic heart valve replacement or structural cardiac abnormality including moderate or severe heart valve disease
* Moderate or severe left atrial dilatation
* Known infiltrative cardiomyopathy
* Known left ventricular systolic dysfunction (ejection fraction <45%)
* Pregnancy
* Co-morbidities known to be associated with an inflammatory response (eg. Rheumatoid arthritis)
* Unexplained baseline elevation of ESR or CRP above the normal lab reference ranges
* Additional ablation lesions beyond pulmonary vein isolation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of recurrence of atrial arrhythmia in the 3 months following ablation | 3 months
  Whether patients have experienced a recurrence of atrial arrhythmia (AF, left atrial flutter or left atrial tachycardia) in the 3 months following their ablation

SECONDARY OUTCOMES:
Rate and degree of rise of inflammatory markers in the 3 months following ablation | 3 months
  Inflammatory blood markers such as CRP
Degree of endothelial dysfunction in the 3 months following ablation (EndoPAT testing) | 3 months
  Endothelial function measured using the EndoPAT technology

CONTACTS AND LOCATIONS:
Overall Officials: Gwilym Morris, BM BCh MRCP PhD, Principal Investigator — The University of Manchester

IPD SHARING:
Plan to Share IPD: No